CLINICAL TRIAL: NCT03193515
Title: A Novel Multiplex ELISA Assay for Surveilling Patients With History of Bladder Cancer
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); University of Texas (Other); University of California, San Francisco (Other); Nonagen Bioscience Corporation (Industry); Kyoto University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Charles Rosser, Professor, Cedars-Sinai Medical Center
Other Study IDs: Rosser-2015-6; R01CA198887 (NIH)
Record Dates: First submitted 2017-06-17; First posted 2017-06-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine collection (minimal 50 mL) and cystoscopy (+ biopsy w/in 4 weeks, if abnormal noted)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Voided urinary cytology (VUC) is the most widely used urine-based assay for detecting bladder cancer (BCa); however, it fails to detect approximately 50% of low-grade or early stage BCa when it is most curable. Furthermore, the detection rate of VUC for recurrent BCa is not much better. Because of this severe limitation, all patients who are under surveillance to monitor for recurrent BCa must undergo an invasive examination of the urinary bladder, where a miniature camera is inserted into the bladder and the bladder inspected (cystoscopy). We propose to improve the non-invasive detection of recurrent BCa by further validating a multiplex ELISA assay directed at a BCa-associated diagnostic signature in voided urine samples.

ELIGIBILITY:
Inclusion Criteria

Participants must be:

* Age 18 years or older
* Have a history of non-muscle invasive bladder cancer or muscle invasive bladder cancer treated by bladder sparing techniques (or not yet treated) and diagnosed within the past 24 months on cystoscopic surveillance
* Participants may be treated with adjuvant intravesical therapy
* Willing and able to give written informed consent (see Appendix 1)
* Be willing to adhere to the surveillance regimen (high risk and intermediate risk seen every 3 months for 2 years; low risk seen every 6-12 months for 2 years)

Exclusion Criteria:

Participants must not:

* Have had radical cystectomy
* History of previous cancer (excluding bladder, basal and squamous cell skin cancer) within the past 3 years
* Have a known active urinary tract infection or urinary retention
* Have active stone disease (renal or bladder) or renal insufficiency (creatinine >2.0 mg/dL) - Serum creatinine value can be up to 60 days before consent, otherwise repeat.
* Have ureteral stents, nephrostomy tubes or bowel interposition
* Have recent genitourinary instrumentation (within 10 days prior to signing consent)
* Be unable or unwilling to complete the surveillance regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of non-muscle invasive bladder cancer or muscle invasive bladder cancer treated by bladder sparing techniques (or not yet treated) and diagnosed within the past 24 months on cystoscopic surveillance
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-12-30 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of multiplex ELISA assay will be confirmed by cystoscopy. | 2 years
  To examine the sensitivity and specificity of the multiplex ELISA assay directed at a BCa-associated diagnostic signature in voided urine samples to reference standard of cystoscopy in a prospective longitudinal cohort of 300 participants with a history of BCa currently on cancer surveillance.

SECONDARY OUTCOMES:
Sensitivity and specificity of multiplex ELISA assay will be compared to VUC and NMP22 BladderCheck. | 2 years
  To compare the sensitivity and specificity of the multiplex ELISA assay to VUC and NMP22® BladderChek to reference standard of cystoscopy in this cohort.
  To develop a BCa risk calculator from this cohort using cutting edge machine learning techniques (e.g., random forest) incorporating biomarker data and clinical data.

CONTACTS AND LOCATIONS:
Overall Officials: Hideki Furuya, PhD, Principal Investigator — Cedars-Sinai Medical Center; Charles Rosser, Study Director — Nonagen Bioscience Corporation
Locations (4):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
- Kyoto University Graduate School of Medicine, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furuya H, Sakatani T, Tanaka S, Murakami K, Waldron RT, Hogrefe W, Rosser CJ. Bladder cancer risk stratification with the Oncuria 10-plex bead-based urinalysis assay using three different Luminex xMAP instrumentation platforms. J Transl Med. 2024 Jan 2;22(1):8. doi: 10.1186/s12967-023-04811-2. PMID 38167321
- [Derived] Furuya H, Sakatani T, Tanaka S, Murakami K, Waldron RT, Hogrefe W, Rosser CJ. Bladder cancer risk stratification with the Oncuria 10-plex bead-based urinalysis assay using three different Luminex xMAP instrumentation platforms. Res Sq [Preprint]. 2023 Nov 25:rs.3.rs-3635581. doi: 10.21203/rs.3.rs-3635581/v1. PMID 38045238